CLINICAL TRIAL: NCT03604822
Title: Measuring the Effects of a Music Therapy Protocol on Respiratory and Bulbar Functions of Patients With Early and Mid-stage Amyotrophic Lateral Sclerosis: Mixed Methods Single Case Study Series
Brief Title: Music Therapy Protocol to Support Bulbar and Respiratory Functions in ALS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alisa Apreleva (Other)
Collaborators: ALS Centre Moscow (Unknown)
Responsible Party: Sponsor-Investigator, Alisa Apreleva, Principal Investigator, Anglia Ruskin University
Organization: Anglia Ruskin University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ALSMT01
Record Dates: First submitted 2018-07-07; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Motor Neuron Disease, Amyotrophic Lateral Sclerosis; ALS (Amyotrophic Lateral Sclerosis); Dysarthria, Flaccid; Dysarthria, Spastic; Dysarthria, Mixed; Dysphagia; Dyspnea; Aspiration Pneumonia; Hypernasality; Breathlessness
Keywords: Music Therapy; Neurologic Music Therapy; Rehabilitation; Amyotrophic Lateral Sclerosis; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Dysarthria; Deglutition Disorders; Dyspnea; Pneumonia, Aspiration | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Single-subject design (Repeated measures)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music therapy protocol (Experimental): Each participant received 12 home-based music therapy treatment sessions over 6-week time period.
  Interventions: Procedure: Music therapy

INTERVENTIONS:
Procedure: Music therapy — ALS-specific, individualized MT protocol was delivered to study participants in their homes twice weekly for the duration of six weeks by the researcher. Facilitating music structures were composed by the researcher to support cueing, timing and intensity of breathing and vocalization exercises. These structures were regularly modified to suit the unique capabilities, current individual demands and progress of each participant. One familiar song, selected by the participant, was used for each participant in therapeutic singing exercise closing each session. Individualized exercises sets for independent practice were provided at session 3 to each participants. ALS-specific voice health guidelines were provided for participants prior to start of the treatment.

SUMMARY:
This study evaluates potential of music therapy treatment to support breathing, speech, swallow and cough of persons with amyotrophic lateral sclerosis (ALS). Music therapy is the clinical use of music and its elements to enhance human health and wellbeing. Application of music therapy principles in neurorehabilitation allow to treat cognitive, sensory, and motor dysfunctions.

DETAILED DESCRIPTION:
ALS clinical presentation and pathophysiology

Amyotrophic lateral sclerosis (ALS) is a group of rapidly progressive fatal neurological diseases involving the brain and spinal cord. Clinical presentation is phenotypically heterogeneous and depends on the type of onset. The pathophysiology mechanisms behind ALS are not clear and may include oxidative stress, protein misfolding and aggregation, skeletal muscle dysfunction, glutamate excitotoxicity, mitochondrial dysfunction, neuroinflammation, and apoptosis. Whilst in the past ALS was considered distinctly a disorder of the motor system, current evidence suggests that some cognitive (ALSci) or behavioural (ALSbi) impairment occurs in up to 50% of cases, and co-morbid dementia (ALS-FTD) occurs in approximately 14% of patients with a new diagnosis of ALS. The notion that "pure" ALS and "pure" FTD may present two extremes of one disease continuum is reinforced by identification of transactive response DNA-binding protein 43 (TDP-43) as a major pathological substrate underlying both diseases. Emotional lability (pseudobulbar affect), a symptom frequently correlated with bulbar involvement in ALS, may also be confusing and disruptive, especially when communicating with those who are not aware of the nature of the problem.

Music therapy potential in multidisciplinary model of ALS care

Considering the multiple and complex needs of people with ALS (PALS), the National Institute for Health and Care Excellence (UK) guideline [NG42] suggests coordinated care using a clinic based, specialist ALS multidisciplinary team approach. American Academy of Neurology recommends multidisciplinary team (MDT) model of care where patients are seen by a comprehensive team of health care professionals who each focus on specific health domains including walking, breathing, speaking, eating, activities of daily living, and psychosocial needs during one clinical visit. Multidisciplinary ALS care has been shown to increase survival of people with PALS and to improve their mental QoL.

More rehabilitation options have to be considered for PALS, enabling them to reach their fullest potential, delaying the disease progression and prolonging lifespan. Music therapy (MT) is the clinical use of music and its elements to accomplish individualized health goals within a therapeutic relationship. Music engages vast network of regions located in both hemispheres of the brain and shares processing components with other functions, such as those involved in language, movement, reasoning and experiencing emotions. Application of MT principles in neurorehabilitation allow to treat cognitive, sensory, and motor dysfunctions. Professionally trained music therapists are well equipped to provide symptomatic care for people with neurodegenerative diseases, adapting to increasing and changing disability of each patient as the disease progresses, whilst maintaining and developing trusting therapeutic relationship established early in the disease course. Albeit currently underused, MT could be one of the modalities of supportive rehabilitation in ALS.

Research on clinical MT applications for ALS is scarce and presents significant challenges due to heterogeneity of ALS clinical presentation and progression, poor scientific understanding of the disease mechanisms and the ethical issues of research involving terminally ill people. It has been suggested that MT could contribute to interdisciplinary ALS care. There is anecdotal evidence that MT increases mind-body connection, reduces distressing physical symptoms such as dyspnoea and pain, and associated feelings of loneliness, anxiety and sadness for patients with advanced ALS, is "pleasant and restorative" for PALS with tracheostomy and their families , and provides families affected by ALS with opportunities for shared meaningful activities. The first randomized controlled trial (RCT) of music therapy effect on people living with ALS found that active MT increased communication, improved QoL and decreased the physical symptoms of the disease for people with ALS during hospital stay. Music-assisted relaxation may be a useful strategy to optimize noninvasive ventilation (NIV) experience for people with ALS.

It may be concluded that, firstly, in most cases, MT is available for PALS at the end of life, when natural communication and motor functions are lost or limited, that music therapists are normally not included into multidisciplinary model of ALS care and that the predominant type of music intervention being used for treatment is music listening. Secondly, little research has been done to understand the effects of MT interventions conducted with patients at earlier stages of ALS and no published research addressing the use of MT techniques for neurorehabilitation (e.g. supporting motor, cognitive, respiratory, swallowing, speech functions) of PALS has been found.

Role of exercise in ALS treatment

Prior to recently the exercise has been discouraged for people with ALS, the recommendation based on the assumption that exercise can lead to muscle fatigue and, hence, increase patient's disability. This assumption however is not supported by scientific evidence, whilst, to the contrary, there is evidence that physical inactivity secondary to ALS may lead to cardiovascular deconditioning, disuse weakness and consequential muscle atrophy. Existing literature reviews support evidence for moderate exercise in ALS, whilst highlighting importance of supervised, individualized training programs. Cochrane review concluded there was no solid evidence to deem exercise in ALS beneficial or harmful and emphasized the need for further research. Recent data suggests that exercise may be beneficial for cellular and morphological adaptations in motor neuron function and thus may help to maintain motor function. Finally, preliminary results of a new RCT suggest that strictly monitored exercise programs reduce motor deterioration in ALS. Thus, in current clinical practice regular moderate exercise is encouraged for people with ALS to prolong mobility and independence.

MT for management of bulbar and respiratory symptoms in ALS

Even more so than in case of the general physical exercise, there is lasting controversy in regards to the role of exercise in management of bulbar and respiratory ALS symptoms. 93% of people with ALS experience speech impairments and 85% present with swallowing dysfunction at some point during the disease progression. Loss of natural communication is regarded by the patients as one of the worst aspects of the disease. Respiratory failure has been cited as the leading cause of death, and weakening of the respiratory function and adherence to NIV as the leading causes of anxiety of people with ALS. Patients with dysphagia reported social isolation, fear and decreased mental health. Dysphagia and malnutrition contribute to 25.9% of ALS mortality and increase the risk of death by 7.7 times. Aspiration pneumonia and dehydration have also been cited among the leading factors contributing to mortality in ALS.

Although there is lack of evidence supporting the use of strengthening exercises for improving speech in patients with ALS, there is no evidence of such exercises being harmful. Respiratory training may have positive effect on respiratory and swallowing functions of people with ALS. Whilst physical and psycho-emotional needs of people with ALS that MT can potentially attend to are many and varied, literature overview and empirical evidence suggest that researching the role of individualized, carefully monitored MT program to support respiratory and bulbar functions of people with ALS currently constitute the highest priority as these functions directly affect survival.

Study aim and significance

Applied MT research in multidisciplinary clinical context allows to systematically look at bulbar and respiratory functions support in ALS, which is important to do, since swallowing, vocalization and breathing are tightly coordinated, and close relationship exists between these processes, in terms of location and activation of the neurons.

This study intends to determine feasibility of a MT protocol as intervention to support respiration, cough, swallowing and speech functions of persons with amyotrophic lateral sclerosis (PALS). Since MT constitutes a new treatment modality for bulbar and respiratory dysfunction in ALS, the study is focused primarily on safety and tolerability of the treatment protocol.

Music therapy treatment protocol

Upper motor neurons and lower motor neurons deterioration in ALS results in dysarthria and dysphagia of spastic-flaccid type, although actual presentation varies in each patient and changes with the disease progression. Generally, lower motor neurone (LMN) involvement, characteristic of bulbar onset, leads to flaccid presentation, whilst degeneration of upper motor neurone (UMN), characteristic of spinal onset, results in spasticity of bulbar muscles. Muscle relaxation and moderate exercise, as well as learning efficient breathing and voice production techniques, voice care techniques and ALS-specific communication strategies may be helpful, rather than rigorous strengthening oral motor exercises. The protocol serves the following primary therapy objectives:

* to increase breath support,
* to increase muscle relaxation,
* to increase speech rate,
* to prevent / decrease hypernasality,
* to maintain swallowing coordination.

ALS-specific, individualized MT protocol was delivered to study participants in their homes twice weekly for the duration of six weeks by the researcher, who is a board certified music therapist and neurologic music therapist, with experience of working with this patient group and in this setting. Facilitating music structures have been composed by the researcher to support cueing, timing and intensity of breathing and vocalization exercises. These structures were regularly modified to suit the unique capabilities, current individual demands and progress of each participant. One familiar song, selected by the participant, was used for each participant in therapeutic singing exercise closing each session.

Data collection

Assessing bulbar dysfunction in ALS presents additional challenge to a researcher, as the existing tools may be not sensitive enough to reliably measure the change, given that ALS is a rapidly degenerating disease and that the rate of deterioration varies greatly from patient to patient. An array of subjective and objective measurements for bulbar and respiratory changes are used, including standard respiratory tools (FVC, MIP, MEP, PCF), videofluoroscopic swallow study, visual analogue scales for ease of speech and respiration, machine analysis of recorded vocal samples, semi-structured interviews and session descriptions, to explore the feasibility of systematic bulbar and respiratory assessment in ALS for future research.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients at ALS Centre Moscow (consecutive sampling)
* Diagnosis of probable or definite ALS by the revised El Escorial criteria confirmed by neurologist at ALS Moscow Centre prior to screening for enrollment.
* Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R) bulbar subscore ≥ 9, but ≤ 11, where bulbar score=the sum of ALSFRS-R questions 1-3 (maximum score of 12)
* Forced vital capacity (FVC) greater than 60%
* Unimpaired cognition as evidenced by Edinburgh Cognitive and Behavioural ALS Screen (ECAS) cut-off scores adjusted for age and education
* Able to consent to treatment
* Native speakers of Russian

Exclusion Criteria:

* Tracheostomy or mechanical ventilation
* Diaphragmatic pacer
* Significant concurrent respiratory disease
* Allergies to barium
* Receiving any other experimental treatment for dysarthria, dysphagia, dystussia and dyspnoea for the duration of the study
* Receiving any other music therapy treatment for the duration of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Change of Forced Vital Capacity (FVC) from baseline at Week 6, Week 12, Week 16 | Throughout the field phase of the study (16 weeks)
  FVC is a standard spirometry test which measures the volume of air that can forcibly be blown out after full inspiration.
Change of Maximal Inspiratory Pressure (MIP) from baseline at Week 6, Week 12, Week 16 | Throughout the field phase of the study (16 weeks)
  MIP is the inspiratory pressure generated against a completely occluded airway; used to evaluate inspiratory respiratory muscle strength.
Change of Maximal Expiratory Pressure (MEP) from baseline at Week 6, Week 12, Week 16 | Throughout the field phase of the study (16 weeks)
  MIP is a measure of the strength of respiratory muscles, obtained by having the patient exhale as strongly as possible against a mouthpiece.
Change of Peak Cough Flow (PCF) from baseline at Week 6, Week 12, Week 16 | Throughout the field phase of the study (16 weeks)
  PCF is a measure of cough effectiveness, portable peak flow meter was used.
Change of Center for Neurologic Study Bulbar Function Scale (CNS-BFS) Swallowing subscore from baseline at Week 6, Week 12, Week 16 | Throughout the field phase of the study (16 weeks)
  The Center for Neurologic Study Bulbar Function Scale (CNS-BFS) consists of three domains (swallowing, speech, and salivation), each of which is assessed with a 7-item, self report questionnaire. Each question is scored from "1" (does not apply) to "5" (applies most of the time). Swallowing domain subscore can range from "7" (best outcome) to "35" (worst outcome).
Change of Center for Neurologic Study Bulbar Function Scale (CNS-BFS) Speech subscore from baseline at Week 6, Week 12, Week 16 | Throughout the field phase of the study (16 weeks)
  The Center for Neurologic Study Bulbar Function Scale (CNS-BFS) consists of three domains (swallowing, speech, and salivation), each of which is assessed with a 7-item, self report questionnaire. Each question is scored from "1" (does not apply) to "5" (applies most of the time). Speech domain subscore can range from "7" (best outcome) to "35" (worst outcome).
Change in video fluoroscopic swallowing study (VFSS) results from baseline at Week 6, Week 12 | Throughout the field phase of the study (16 weeks)
  VFSS is an x-ray-based method of evaluating a person's swallowing ability.
Change in acoustic assessment parameters of recorded voice from baseline at Week 6, Week 12, Week 16 | Throughout the field phase of the study (16 weeks)
  Machine-analyzed set of structured voice samples.
Change in Visual Analogue Scale for current perceived ease of respiration from pre-treatment to post-treatment | Throughout the therapy phase (6 weeks)
  Visual Analogue Scale (VAS) for current perceived ease of respiration is a one question 10-point scale administered at the beginning and at the end of every music therapy session to assess short-term change in current perceived ease of respiration. The outcome can range from "1" (very difficult) to "10" (very easy).
Change of Visual Analogue Scale for current perceived ease of speech from pre-treatment to post-treatment | Throughout the therapy phase (6 weeks)
  Visual Analogue Scale (VAS) for current perceived ease of speech is a one question 10-point scale administered at the beginning and at the end of every music therapy session to assess short-term change in current perceived ease of speech. The outcome can range from "1" (very difficult) to "10" (very easy).
Phenomenological analysis of participant semi-structured interviews pre-treatment | Week 5
  Analysis of participant's answers to open questions in regards to expectations for music therapy treatment
Phenomenological analysis of caregiver semi-structured interview pre-treatment | Week 5
  Analysis of main caregiver's answers to open questions in regards to expectations for music therapy treatment
Phenomenological analysis of treatment sessions documentation | Throughout the therapy phase (6 weeks)
  Analysis of narrative accounts of music therapy sessions submitted by the therapist
Phenomenological analysis of participant semi-structured interviews post-treatment | Week 13
  Analysis of participant's answers to open questions in regards to impressions of music therapy treatment
Phenomenological analysis of caregiver semi-structured interview post-treatment | Week 13
  Analysis of main caregiver's answers to open questions in regards to impressions of music therapy treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alisa Apreleva, MA, Principal Investigator — Anglia Ruskin University
Locations (2):
- ALS Moscow Centre, Moscow, Russia
- Cambridge Institute for Music Therapy Research (CIMTR), Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymized individual participant data for all outcome measures will be made available.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Within 6 months of study completion, indefinitely.
Access Criteria: Contact sponsor-investigator for data access.
URL: http://alsmusictherapy.org

REFERENCES:
- [Background] de Almeida JP, Silvestre R, Pinto AC, de Carvalho M. Exercise and amyotrophic lateral sclerosis. Neurol Sci. 2012 Feb;33(1):9-15. doi: 10.1007/s10072-011-0921-9. Epub 2012 Jan 7. PMID 22228269
- [Background] Andersen PM, Borasio GD, Dengler R, Hardiman O, Kollewe K, Leigh PN, Pradat PF, Silani V, Tomik B; EFNS Task Force on Diagnosis and Management of Amyotrophic Lateral Sclerosis. EFNS task force on management of amyotrophic lateral sclerosis: guidelines for diagnosing and clinical care of patients and relatives. Eur J Neurol. 2005 Dec;12(12):921-38. doi: 10.1111/j.1468-1331.2005.01351.x. PMID 16324086
- [Background] Ashworth NL, Satkunam LE, Deforge D. Treatment for spasticity in amyotrophic lateral sclerosis/motor neuron disease. Cochrane Database Syst Rev. 2012 Feb 15;2012(2):CD004156. doi: 10.1002/14651858.CD004156.pub4. PMID 22336799
- [Background] Baker F, Wigram T, Gold C. The effects of a song-singing programme on the affective speaking intonation of people with traumatic brain injury. Brain Inj. 2005 Jul;19(7):519-28. doi: 10.1080/02699050400005150. PMID 16134740
- [Background] Bello-Haas VD, Florence JM, Kloos AD, Scheirbecker J, Lopate G, Hayes SM, Pioro EP, Mitsumoto H. A randomized controlled trial of resistance exercise in individuals with ALS. Neurology. 2007 Jun 5;68(23):2003-7. doi: 10.1212/01.wnl.0000264418.92308.a4. PMID 17548549
- [Background] Beukelman D, Fager S, Nordness A. Communication Support for People with ALS. Neurol Res Int. 2011;2011:714693. doi: 10.1155/2011/714693. Epub 2011 Apr 14. PMID 21603029
- [Background] Bonafede R, Mariotti R. ALS Pathogenesis and Therapeutic Approaches: The Role of Mesenchymal Stem Cells and Extracellular Vesicles. Front Cell Neurosci. 2017 Mar 21;11:80. doi: 10.3389/fncel.2017.00080. eCollection 2017. PMID 28377696
- [Background] Bowen LK, Hands GL, Pradhan S, Stepp CE. Effects of Parkinson's Disease on Fundamental Frequency Variability in Running Speech. J Med Speech Lang Pathol. 2013 Sep;21(3):235-244. PMID 25838754
- [Background] Bredart A, Marrel A, Abetz-Webb L, Lasch K, Acquadro C. Interviewing to develop Patient-Reported Outcome (PRO) measures for clinical research: eliciting patients' experience. Health Qual Life Outcomes. 2014 Feb 5;12:15. doi: 10.1186/1477-7525-12-15. PMID 24499454
- [Background] Bukowska AA, Krezalek P, Mirek E, Bujas P, Marchewka A. Neurologic Music Therapy Training for Mobility and Stability Rehabilitation with Parkinson's Disease - A Pilot Study. Front Hum Neurosci. 2016 Jan 26;9:710. doi: 10.3389/fnhum.2015.00710. eCollection 2015. PMID 26858628
- [Background] Chen A, Montes J, Mitsumoto H. The role of exercise in amyotrophic lateral sclerosis. Phys Med Rehabil Clin N Am. 2008 Aug;19(3):545-57, ix-x. doi: 10.1016/j.pmr.2008.02.003. PMID 18625415
- [Background] Chiao GZ, Larson CR, Yajima Y, Ko P, Kahrilas PJ. Neuronal activity in nucleus ambiguous during deglutition and vocalization in conscious monkeys. Exp Brain Res. 1994;100(1):29-38. doi: 10.1007/BF00227276. PMID 7813650
- [Background] Chio A, Logroscino G, Hardiman O, Swingler R, Mitchell D, Beghi E, Traynor BG; Eurals Consortium. Prognostic factors in ALS: A critical review. Amyotroph Lateral Scler. 2009 Oct-Dec;10(5-6):310-23. doi: 10.3109/17482960802566824. PMID 19922118
- [Background] Cohen, N. S. 1992. The effect of singing instruction on the speech production of neurologically impaired persons. Journal of Music Therapy, 29(87-103)
- [Background] Czaplinski A, Yen AA, Appel SH. Forced vital capacity (FVC) as an indicator of survival and disease progression in an ALS clinic population. J Neurol Neurosurg Psychiatry. 2006 Mar;77(3):390-2. doi: 10.1136/jnnp.2005.072660. PMID 16484652
- [Background] Davies, R., Baker, F. A., Tamplin, J., Bajo, E., Bolger, K., Sheers, N. & Berlowitz, D. 2016. Music-assisted relaxation during transition to non-invasive ventilation in people with motor neuron disease: A qualitative case series. British Journal of Music Therapy, 30(2), pp 74-82.
- [Background] Donovan NJ, Kendall DL, Young ME, Rosenbek JC. The communicative effectiveness survey: preliminary evidence of construct validity. Am J Speech Lang Pathol. 2008 Nov;17(4):335-47. doi: 10.1044/1058-0360(2008/07-0010). PMID 18957572
- [Background] Drory VE, Goltsman E, Reznik JG, Mosek A, Korczyn AD. The value of muscle exercise in patients with amyotrophic lateral sclerosis. J Neurol Sci. 2001 Oct 15;191(1-2):133-7. doi: 10.1016/s0022-510x(01)00610-4. PMID 11677004
- [Background] Forrest, L. Using Music Therapy in the Symptom Management of Patients with Motor Neurone Disease. 10th World congress on music therapy, 2002 Oxford, UK.
- [Background] Green JR, Yunusova Y, Kuruvilla MS, Wang J, Pattee GL, Synhorst L, Zinman L, Berry JD. Bulbar and speech motor assessment in ALS: challenges and future directions. Amyotroph Lateral Scler Frontotemporal Degener. 2013 Dec;14(7-8):494-500. doi: 10.3109/21678421.2013.817585. Epub 2013 Jul 30. PMID 23898888
- [Background] Gregory D. Music listening for maintaining attention of older adults with cognitive impairments. J Music Ther. 2002 Winter;39(4):244-64. doi: 10.1093/jmt/39.4.244. PMID 12597728
- [Background] Haneishi E. Effects of a music therapy voice protocol on speech intelligibility, vocal acoustic measures, and mood of individuals with Parkinson's disease. J Music Ther. 2001 Winter;38(4):273-90. doi: 10.1093/jmt/38.4.273. PMID 11796078
- [Background] Hardiman O, Figlewicz DA. The expansions of ALS. Neurology. 2012 Aug 28;79(9):842-3. doi: 10.1212/WNL.0b013e3182662031. Epub 2012 Jul 25. No abstract available. PMID 22843260
- [Background] Hecht M, Hillemacher T, Grasel E, Tigges S, Winterholler M, Heuss D, Hilz MJ, Neundorfer B. Subjective experience and coping in ALS. Amyotroph Lateral Scler Other Motor Neuron Disord. 2002 Dec;3(4):225-31. doi: 10.1080/146608202760839009. PMID 12710513
- [Background] Horne-Thompson A, Grocke D. The effect of music therapy on anxiety in patients who are terminally ill. J Palliat Med. 2008 May;11(4):582-90. doi: 10.1089/jpm.2007.0193. PMID 18454611
- [Background] Jensen L, Djurtoft JB, Bech RD, Nielsen JL, Jorgensen LH, Schroder HD, Frandsen U, Aagaard P, Hvid LG. Influence of Resistance Training on Neuromuscular Function and Physical Capacity in ALS Patients. J Neurodegener Dis. 2017;2017:1436519. doi: 10.1155/2017/1436519. Epub 2017 May 17. PMID 28596929
- [Background] K. Hanson, E., M. Yorkston, K. & Britton, D. 2011. Dysarthria in amyotrophic lateral sclerosis: a systematic review of characteristics, speech treatment, and augmentative and alternative communication options.(Report). Journal of Medical Speech - Language Pathology, 19(3), pp 12
- [Background] Kaub-Wittemer D, Steinbuchel Nv, Wasner M, Laier-Groeneveld G, Borasio GD. Quality of life and psychosocial issues in ventilated patients with amyotrophic lateral sclerosis and their caregivers. J Pain Symptom Manage. 2003 Oct;26(4):890-6. doi: 10.1016/s0885-3924(03)00323-3. PMID 14527757
- [Background] Kim SJ. Music therapy protocol development to enhance swallowing training for stroke patients with dysphagia. J Music Ther. 2010 Summer;47(2):102-19. doi: 10.1093/jmt/47.2.102. PMID 21141768
- [Background] Koelsch S. Brain correlates of music-evoked emotions. Nat Rev Neurosci. 2014 Mar;15(3):170-80. doi: 10.1038/nrn3666. PMID 24552785
- [Background] Kondo, K. 2017. Music therapy for patients with amyotrophic lateral sclerosis receiving home mechanical ventilation. Journal of the Neurological Sciences, 381(561 - 756)
- [Background] Lee J, Littlejohn MA, Simmons Z. Acoustic and tongue kinematic vowel space in speakers with and without dysarthria. Int J Speech Lang Pathol. 2017 Apr;19(2):195-204. doi: 10.1080/17549507.2016.1193899. Epub 2016 Jun 23. PMID 27336197
- [Background] Lings, J. 2014. From 'can't' to 'can' : an exploration of the experience of improvisation with a client with Motor Neurone Disease Counterpoints: Music Therapy Practice in the 21st Century, First BAMT conference. Birmingham, UK
- [Background] Lisle S, Tennison M. Amyotrophic lateral sclerosis: the role of exercise. Curr Sports Med Rep. 2015 Jan;14(1):45-6. doi: 10.1249/JSR.0000000000000122. PMID 25574882
- [Background] Lunetta C, Lizio A, Sansone VA, Cellotto NM, Maestri E, Bettinelli M, Gatti V, Melazzini MG, Meola G, Corbo M. Strictly monitored exercise programs reduce motor deterioration in ALS: preliminary results of a randomized controlled trial. J Neurol. 2016 Jan;263(1):52-60. doi: 10.1007/s00415-015-7924-z. PMID 26477027
- [Background] Magee, W. 1998. Singing my life, playing my self: investigating the use of familiar pre-composed music and unfamiliar improvised music in clinical music therapy with individuals with chronic neurological illness. ProQuest Dissertations Publishing
- [Background] Majmudar S, Wu J, Paganoni S. Rehabilitation in amyotrophic lateral sclerosis: why it matters. Muscle Nerve. 2014 Jul;50(1):4-13. doi: 10.1002/mus.24202. Epub 2014 May 17. PMID 24510737
- [Background] Matsuo K, Palmer JB. Coordination of Mastication, Swallowing and Breathing. Jpn Dent Sci Rev. 2009 May 1;45(1):31-40. doi: 10.1016/j.jdsr.2009.03.004. PMID 20161022
- [Background] McCullough GH, Kamarunas E, Mann GC, Schmidley JW, Robbins JA, Crary MA. Effects of Mendelsohn maneuver on measures of swallowing duration post stroke. Top Stroke Rehabil. 2012 May-Jun;19(3):234-43. doi: 10.1310/tsr1903-234. PMID 22668678
- [Background] Mefferd AS, Green JR, Pattee G. A novel fixed-target task to determine articulatory speed constraints in persons with amyotrophic lateral sclerosis. J Commun Disord. 2012 Jan-Feb;45(1):35-45. doi: 10.1016/j.jcomdis.2011.09.002. Epub 2011 Sep 28. PMID 22000045
- [Background] Mendelsohn MS, McConnel FM. Function in the pharyngoesophageal segment. Laryngoscope. 1987 Apr;97(4):483-9. doi: 10.1288/00005537-198704000-00014. PMID 3561135
- [Background] Miller RG, Jackson CE, Kasarskis EJ, England JD, Forshew D, Johnston W, Kalra S, Katz JS, Mitsumoto H, Rosenfeld J, Shoesmith C, Strong MJ, Woolley SC; Quality Standards Subcommittee of the American Academy of Neurology. Practice parameter update: the care of the patient with amyotrophic lateral sclerosis: multidisciplinary care, symptom management, and cognitive/behavioral impairment (an evidence-based review): report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2009 Oct 13;73(15):1227-33. doi: 10.1212/WNL.0b013e3181bc01a4. PMID 19822873
- [Background] Nishio, M. & Niimi, S. 2000. Changes over Time in Dysarthric Patients with Amyotrophic Lateral Sclerosis (ALS): A Study of Changes in Speaking Rate and Maximum Repetition Rate (MRR). Clinical Linguistics & Phonetics, 14(7), pp 485-497
- [Background] Oh SI, Park A, Kim HJ, Oh KW, Choi H, Kwon MJ, Ki CS, Kim HT, Kim SH. Spectrum of cognitive impairment in Korean ALS patients without known genetic mutations. PLoS One. 2014 Feb 3;9(2):e87163. doi: 10.1371/journal.pone.0087163. eCollection 2014. PMID 24498297
- [Background] Paganoni S, Karam C, Joyce N, Bedlack R, Carter GT. Comprehensive rehabilitative care across the spectrum of amyotrophic lateral sclerosis. NeuroRehabilitation. 2015;37(1):53-68. doi: 10.3233/NRE-151240. PMID 26409693
- [Background] Palovcak M, Mancinelli JM, Elman LB, McCluskey L. Diagnostic and therapeutic methods in the management of dysphagia in the ALS population: issues in efficacy for the out-patient setting. NeuroRehabilitation. 2007;22(6):417-23. PMID 18198426
- [Background] Paris G, Martinaud O, Petit A, Cuvelier A, Hannequin D, Roppeneck P, Verin E. Oropharyngeal dysphagia in amyotrophic lateral sclerosis alters quality of life. J Oral Rehabil. 2013 Mar;40(3):199-204. doi: 10.1111/joor.12019. Epub 2012 Dec 27. PMID 23278936
- [Background] Patel BP, Hamadeh MJ. Nutritional and exercise-based interventions in the treatment of amyotrophic lateral sclerosis. Clin Nutr. 2009 Dec;28(6):604-17. doi: 10.1016/j.clnu.2009.06.002. Epub 2009 Sep 25. PMID 19782443
- [Background] Peretz I, Zatorre RJ. Brain organization for music processing. Annu Rev Psychol. 2005;56:89-114. doi: 10.1146/annurev.psych.56.091103.070225. PMID 15709930
- [Background] Petering, H. 2005. Fostering hope through music therapy with people with Motor Neurone Disease 11th World Congress of Music Therapy, Brisbane, Australia
- [Background] Phukan J, Elamin M, Bede P, Jordan N, Gallagher L, Byrne S, Lynch C, Pender N, Hardiman O. The syndrome of cognitive impairment in amyotrophic lateral sclerosis: a population-based study. J Neurol Neurosurg Psychiatry. 2012 Jan;83(1):102-8. doi: 10.1136/jnnp-2011-300188. Epub 2011 Aug 11. PMID 21836033
- [Background] Pietkiewicz, I. & Smith, J. A. 2014. A practical guide to using Interpretative Phenomenological Analysis in qualitative research psychology. Czasopismo Psychologiczne - Psychological Journal, 20(1), pp 7 - 14
- [Background] Pinto AC, Alves M, Nogueira A, Evangelista T, Carvalho J, Coelho A, de Carvalho M, Sales-Luis ML. Can amyotrophic lateral sclerosis patients with respiratory insufficiency exercise? J Neurol Sci. 1999 Oct 31;169(1-2):69-75. doi: 10.1016/s0022-510x(99)00218-x. PMID 10540010
- [Background] Pinto S, de Carvalho M. Correlation between Forced Vital Capacity and Slow Vital Capacity for the assessment of respiratory involvement in Amyotrophic Lateral Sclerosis: a prospective study. Amyotroph Lateral Scler Frontotemporal Degener. 2017 Feb;18(1-2):86-91. doi: 10.1080/21678421.2016.1249486. Epub 2016 Dec 4. PMID 27915482
- [Background] Pinto S, Swash M, de Carvalho M. Respiratory exercise in amyotrophic lateral sclerosis. Amyotroph Lateral Scler. 2012 Jan;13(1):33-43. doi: 10.3109/17482968.2011.626052. PMID 22214352
- [Background] Plowman EK. Is There a Role for Exercise in the Management of Bulbar Dysfunction in Amyotrophic Lateral Sclerosis? J Speech Lang Hear Res. 2015 Aug 1;58(4):1151-66. doi: 10.1044/2015_JSLHR-S-14-0270. PMID 26091205
- [Background] Plowman EK, Tabor LC, Robison R, Gaziano J, Dion C, Watts SA, Vu T, Gooch C. Discriminant ability of the Eating Assessment Tool-10 to detect aspiration in individuals with amyotrophic lateral sclerosis. Neurogastroenterol Motil. 2016 Jan;28(1):85-90. doi: 10.1111/nmo.12700. Epub 2015 Oct 28. PMID 26510823
- [Background] Plowman EK, Watts SA, Tabor L, Robison R, Gaziano J, Domer AS, Richter J, Vu T, Gooch C. Impact of expiratory strength training in amyotrophic lateral sclerosis. Muscle Nerve. 2016 Jun;54(1):48-53. doi: 10.1002/mus.24990. Epub 2016 Mar 3. PMID 26599236
- [Background] Qureshi MM, Hayden D, Urbinelli L, Ferrante K, Newhall K, Myers D, Hilgenberg S, Smart R, Brown RH, Cudkowicz ME. Analysis of factors that modify susceptibility and rate of progression in amyotrophic lateral sclerosis (ALS). Amyotroph Lateral Scler. 2006 Sep;7(3):173-82. doi: 10.1080/14660820600640596. PMID 16963407
- [Background] Raglio A, Bellelli G, Traficante D, Gianotti M, Ubezio MC, Villani D, Trabucchi M. Efficacy of music therapy in the treatment of behavioral and psychiatric symptoms of dementia. Alzheimer Dis Assoc Disord. 2008 Apr-Jun;22(2):158-62. doi: 10.1097/WAD.0b013e3181630b6f. PMID 18525288
- [Background] Ramig LA, Scherer RC, Titze IR, Ringel SP. Acoustic analysis of voices of patients with neurologic disease: rationale and preliminary data. Ann Otol Rhinol Laryngol. 1988 Mar-Apr;97(2 Pt 1):164-72. doi: 10.1177/000348948809700214. PMID 2965542
- [Background] Zatorre RJ, Chen JL, Penhune VB. When the brain plays music: auditory-motor interactions in music perception and production. Nat Rev Neurosci. 2007 Jul;8(7):547-58. doi: 10.1038/nrn2152. PMID 17585307
- [Background] Rong P, Yunusova Y, Wang J, Zinman L, Pattee GL, Berry JD, Perry B, Green JR. Predicting Speech Intelligibility Decline in Amyotrophic Lateral Sclerosis Based on the Deterioration of Individual Speech Subsystems. PLoS One. 2016 May 5;11(5):e0154971. doi: 10.1371/journal.pone.0154971. eCollection 2016. PMID 27148967
- [Background] Rooney J, Burke T, Vajda A, Heverin M, Hardiman O. What does the ALSFRS-R really measure? A longitudinal and survival analysis of functional dimension subscores in amyotrophic lateral sclerosis. J Neurol Neurosurg Psychiatry. 2017 May;88(5):381-385. doi: 10.1136/jnnp-2016-314661. Epub 2016 Nov 25. PMID 27888187
- [Background] Schmid, W. 2016. MusicALS: home-based music therapy for individuals with amyotrophic lateral sclerosis (ALS) and their caring families. Nord. J. Music Ther., 25(sup1), pp 66-66
- [Background] Sinaki M, Mulder DW. Amyotrophic lateral sclerosis: relationship between serum creatine kinase level and patient survival. Arch Phys Med Rehabil. 1986 Mar;67(3):169-71. doi: 10.1016/0003-9993(86)90064-x. PMID 3954579
- [Background] Strand EA, Buder EH, Yorkston KM, Ramig LO. Differential phonatory characteristics of four women with amyotrophic lateral sclerosis. J Voice. 1994 Dec;8(4):327-39. doi: 10.1016/s0892-1997(05)80281-4. PMID 7858668
- [Background] Sarkamo T, Tervaniemi M, Laitinen S, Forsblom A, Soinila S, Mikkonen M, Autti T, Silvennoinen HM, Erkkila J, Laine M, Peretz I, Hietanen M. Music listening enhances cognitive recovery and mood after middle cerebral artery stroke. Brain. 2008 Mar;131(Pt 3):866-76. doi: 10.1093/brain/awn013. PMID 18287122
- [Background] Tabor LC, Rosado KM, Robison R, Hegland K, Humbert IA, Plowman EK. Respiratory training in an individual with amyotrophic lateral sclerosis. Ann Clin Transl Neurol. 2016 Sep 1;3(10):819-823. doi: 10.1002/acn3.342. eCollection 2016 Oct. PMID 27752517
- [Background] Tamplin J. A pilot study into the effect of vocal exercises and singing on dysarthric speech. NeuroRehabilitation. 2008;23(3):207-16. PMID 18560137
- [Background] Tamplin, J. & Grocke, D. 2008. A Music Therapy Treatment Protocol for Acquired Dysarthria Rehabilitation. Music Therapy Perspectives, 26(1), pp 23-29
- [Background] Thaut, M. & H©œmberg, V. 2016. Handbook of neurologic music therapy: Oxford : Oxford University Press
- [Background] Thaut MH, McIntosh GC, Hoemberg V. Neurobiological foundations of neurologic music therapy: rhythmic entrainment and the motor system. Front Psychol. 2015 Feb 18;5:1185. doi: 10.3389/fpsyg.2014.01185. eCollection 2014. PMID 25774137
- [Background] Touré-Tillery, M. & Fishbach, A. 2014. How to Measure Motivation: A Guide for the Experimental Social Psychologist. Social and Personality Psychology Compass, 8(7), pp 328-341
- [Background] Van den Berg JP, Kalmijn S, Lindeman E, Veldink JH, de Visser M, Van der Graaff MM, Wokke JH, Van den Berg LH. Multidisciplinary ALS care improves quality of life in patients with ALS. Neurology. 2005 Oct 25;65(8):1264-7. doi: 10.1212/01.wnl.0000180717.29273.12. PMID 16247055
- [Background] Wiens ME, Reimer MA, Guyn HL. Music therapy as a treatment method for improving respiratory muscle strength in patients with advanced multiple sclerosis: a pilot study. Rehabil Nurs. 1999 Mar-Apr;24(2):74-80. doi: 10.1002/j.2048-7940.1999.tb01840.x. PMID 10410058
- [Background] Wolf J, Safer A, Wohrle JC, Palm F, Nix WA, Maschke M, Grau AJ. [Causes of death in amyotrophic lateral sclerosis : Results from the Rhineland-Palatinate ALS registry]. Nervenarzt. 2017 Aug;88(8):911-918. doi: 10.1007/s00115-017-0293-3. German. PMID 28184974
- [Background] Woo AS. Velopharyngeal dysfunction. Semin Plast Surg. 2012 Nov;26(4):170-7. doi: 10.1055/s-0033-1333882. PMID 24179450
- [Background] Yang R, Huang R, Chen D, Song W, Zeng Y, Zhao B, Zhou D, Shang HF. Causes and places of death of patients with amyotrophic lateral sclerosis in south-west China. Amyotroph Lateral Scler. 2011 May;12(3):206-9. doi: 10.3109/17482968.2011.572979. Epub 2011 Apr 21. PMID 21506897
- [Background] Yunusova Y, Green JR, Wang J, Pattee G, Zinman L. A protocol for comprehensive assessment of bulbar dysfunction in amyotrophic lateral sclerosis (ALS). J Vis Exp. 2011 Feb 21;(48):2422. doi: 10.3791/2422. PMID 21372794
- See also: Cambridge Institute for Music Therapy Research (CIMTR), Anglia Ruskin University — https://www.anglia.ac.uk/cambridge-institute-for-music-therapy-research
- See also: ALS Centre Moscow — https://alsfund.ru/en/